CLINICAL TRIAL: NCT06585969
Title: A Randomised Trial Comparing Trastuzumab Deruxtecan to CDK4/6 Inhibitors in Non-luminal A, ER-positive/HER2-low Metastatic Breast Cancer
Acronym: DISCORDANT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Danish Breast Cancer Cooperative Group (Other)
Responsible Party: Principal Investigator, Tobias Berg, MD, Danish Breast Cancer Cooperative Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DBCG-R25-DISCORDANT
Record Dates: First submitted 2024-08-23; First posted 2024-09-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Breast Cancer; ER-positive Breast Cancer; Luminal B; Her2 Enriched; Basal Like
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan; ribociclib; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Trastuzumab-deruxtecan (Experimental): Trastuzumab deruxtecan until progression or intolerable toxicity: 5.4 mg/kg intravenous on day 1 of a 21 days cycle.
  Interventions: Drug: Trastuzumab deruxtecan (T-DXd)
- Immunohistochemistry guided treatment (standard) (Active Comparator): - CDK4/6 inhibitor with an endocrine therapy until progression og intolerable toxicity
  * CDK4/6 inhibitor: Physician's choice of ribociclib (600mg daily for 21 days in a 4 week schedule) or abemaciclib (125mg twice daily).
  * Endocrine therapy: letrozole (2.5mg daily), anastrozole (1mg daily), exemestane (25mg daily), tamoxifen (20mg daily) or fulvestrant (intramuscular 500mg every 4 weeks)
  Interventions: Drug: Ribociclib with ET; Drug: Abemaciclib with ET

INTERVENTIONS:
Drug: Trastuzumab deruxtecan (T-DXd) — Trastuzumab deruxtexan every three weeks
  Other Names: Enhertu
  Arms: Trastuzumab-deruxtecan
Drug: Ribociclib with ET — Ribociclib with endocrine therapy
  Arms: Immunohistochemistry guided treatment (standard)
Drug: Abemaciclib with ET — Abemaciclib with endocrine therapy
  Arms: Immunohistochemistry guided treatment (standard)

SUMMARY:
The objective of this trial, DBCG R25, will be to evaluate the effect of trastuzumab-deruxtecan versus standard of care on progression-free survival (PFS) in first-line for patients with non-Luminal A, ER-positive/HER2-negative metastatic breast cancer

DETAILED DESCRIPTION:
Study design and setting We will conduct an international, multicentre, open-label, randomised controlled trial. All oncological departments who treat patients with metastatic breast cancer can participate. The EU Clinical Trial Regulation will be applied.

Interventions Trial participants will be randomised to trastuzumab deruxtecan or standard treatment.

Trastuzumab deruxtecan

Patients randomised to trastuzumab deruxtecan will be treated as:

Trastuzumab deruxtecan until progression or intolerable toxicity, Trastuzumab deruxtecan: 5.4 mg/kg intravenous on day 1 of a 21 days cycle.

Standard

Patients randomised to standard will be treated as:

CDK4/6 inhibitor with an endocrine therapy until progression or intolerable toxicity CDK4/6 inhibitor: Physician's choice of ribociclib (600mg daily for 21 days in a 28 days cycle) or abemaciclib (150mg twice daily).

Endocrine therapy: letrozole (2.5mg daily), anastrozole (1mg daily), exemestane (25mg daily), tamoxifen (20mg daily) or fulvestrant (intramuscular 500mg every 4 weeks)

Other treatment Prophylactic antiemetics are allowed, including corticosteroids. Prophylactic antibiotics are allowed if deemed necessary for the patient. G-CSF is allowed when needed.

All other symptomatic treatment to perform best of care is allowed as long as name, administration and length is documented in the chart. Bone targeted agents are allowed. No other antineoplastic treatment is allowed.

Radiological evaluation Patients will initially be scanned every 9-12 weeks as per investigator's or co-investigator's discretion with minimum a CT of the thorax and abdomen or a FDG-PET/CT. Patients with response can have this interval extended. Upon progression treatment/control is to be done according to department preferences, but subsequent treatment and day of death must be registered.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or above.
* Radiologically/pathologically verified metastatic breast cancer.
* ER-positive (1% or more) and HER2-low (HER2 1+ or HER2 2+/ISH-neg)10,11.
* PAM50 Luminal B, HER2-enriched or Basal-like.
* Performance status 0-1.
* Evaluable disease

Exclusion Criteria:

* Patients who are incapable of understanding the written material received
* Patients with inaccessible tumour tissue
* Other malignant disease within 5 years (in situ cervix and non-melanoma skin cancer excluded)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome | Up to 4 years after inclusion
  Progression-free survival (ITT)

SECONDARY OUTCOMES:
Overall survival | Up to 4 years after inclusion
  Overall survival in ITT cohort
PFS by subtype | Up to 4 years after inclusion
  PFS by subtype (Luminal B, HER2-enriched and Basal-like)
OS by subtype | Up to 4 years after inclusion
  OS by subtype (Luminal B, HER2-enriched and Basal-like)
Quality of life | During treatment, estimated 18-24 months
  Quality of life EORTC QLQ-C30/BR23 during treatment and at progression.
Toxicity | During treatment, estimated 18-24 months
  Toxicity on treatment (NCI-CTC v. 5.0)

IPD SHARING:
Plan to Share IPD: Undecided